CLINICAL TRIAL: NCT02485886
Title: Safety and Diagnostic Performance of 68Ga-BMV101 PET/CT in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: 68Ga-BMV101 PET/CT in Patients With Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM09
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2015-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: PET; interstitial pulmonary fibrosis (IPF); cysteine cathepsins; macrophage
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BMV101 injection and PET/CT scan (Experimental): The patients were intravenously injected with 68Ga-BMV101 and underwent PET/CT scan 1 h and 2.5 h after that.
  Interventions: Drug: 68Ga-BMV101

INTERVENTIONS:
Drug: 68Ga-BMV101 — 68Ga-BMV101 were intravenously injected into the patients 1 h before the PET/CT scans.
  Other Names: BMV101 imaging

SUMMARY:
Inflammation mediated by macrophage infiltration plays a vital role in a diverse range of physiological conditions. In particular, recent evidence suggests this type of macrophage response is important for the disease pathology of pulmonary fibrosis. Because cysteine cathepsins are proteases that are highly expressed in antigen presenting cells such as macrophages, they serve as promising biomarkers. Employing non-invasive imaging agents 68Ga-BMV101 that specifically recognize cysteine proteases in immune cells has the potential to not only aid early detection but also significantly aid efforts to monitor progression and patient response to therapy.

DETAILED DESCRIPTION:
For interests in clinical translation of 68Ga-BMV101, an open-label dynamic whole-body PET/CT study was designed to investigate safety and diagnostic performance of 68Ga-BMV101 in patients with idiopathic pulmonary fibrosis (IPF). A single dose of nearly 111 MBq 68Ga-BMV101 will be intravenously injected into healthy volunteers and patients with suspected IPF. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with idiopathic pulmonary fibrosis

* Males and females, ≥18 years old
* Characteristic clinical signs, symptoms and laboratory tests suggesting the diagnosis of IPF.
* The diagnosis of IPF is based on The Centres for Disease Control and Prevention (CDC) criteria for diagnosing IPF. They rely on a combination of clinical, radiological, operative and histological findings, in addition to results of other laboratory tests.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment of lesions | 1 year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of lungs will be measured.

SECONDARY OUTCOMES:
Blood pressure | 24 hours
  Blood pressure of patients will be measured at three time points: right before injection, after scanning, and 24 hours after treatment.
Pulse | 24 hours
  Pulse will be measured at three time points for each patients: right before injection, after scanning, and 24 hours after treatment.
Respiration frequency | 24 hours
  Respiration frequency will be measured at three time points for each patients: right before injection, after scanning, and 24 hours after treatment.
Temperature | 24 hours
  Temperature will be measured at three time points for each patients: right before injection, after scanning, and 24 hours after treatment.
Routine blood test | 24 hours
  Routine blood test of patients will be measured at two time points: right before injection and 24 hours after treatment.
Routine urine test | 24 hours
  Routine urine test of patients will be measured at two time points: right before injection and 24 hours after treatment.
Serum alanine aminotransferase | 24 hours
  Serum alanine aminotransferase of patients will be measured at two time points: right before injection and 24 hours after treatment.
Serum albumin | 24 hours
  Serum albumin of patients will be measured at two time points: right before injection and 24 hours after treatment.
Serum creatinine | 24 hours
  Serum creatinine of patients will be measured at two time points: right before injection and 24 hours after treatment.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of patients and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No